CLINICAL TRIAL: NCT05051683
Title: Combined Endoscopic & Radiologic Intervention For Management Of Acute Perforated Peptic Ulcer : A Randomized Controlled Trial
Brief Title: Combined Endoscopic & Radiologic Intervention For Management Of Acute Perforated Peptic Ulcer
Acronym: ppu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Said Mohamed Said Abdou Negm, lecturer of general surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zagazig General Surgery
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Abdomen, Acute
Keywords: perforated peptic ulcer
MeSH Terms: conditions — Abdomen, Acute; Peptic Ulcer Perforation

STUDY DESIGN:
Intervention Model Description: The investigators included all patients who were developed acute perforated peptic ulcer manifestations and were admitted to our hospital between December 2019 to August 2021. the calculated sample size equal 100 patients divided into two equal groups. Group (1) included 50 patients managed by combined endoscopic & radiologic intervention , group (2) included 50 patients managed by surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (1) (Active Comparator): combined endoscopic & radiologic intervention for management of acute perforated peptic ulcer
  Interventions: Procedure: combined endoscopic & radiologic intervention for management of acute perforated peptic ulcer
- group (2) (No Intervention): surgical management of acute perforated peptic ulcer

INTERVENTIONS:
Procedure: combined endoscopic & radiologic intervention for management of acute perforated peptic ulcer — endoscopic management using stent , clipping and sewing combined with radiologic interventional drainage was used. For duodenal ulcer only metallic stent was used due to narrow space while for gastric ulcer either stent , clipping and sewing were used due to capacious space.
  Arms: group (1)

SUMMARY:
The investigators included all patients who were developed acute perforated peptic ulcer manifestations and were admitted to our hospital between December 2019 to August 2021. The study was approved by the research and Ethics committee of our university and performed in accordance with the code of ethics of the world medical association (Declaration of Helsinki) for studies involving humans. A written informed consent was obtained from all participants. The sample size was calculated using open Epi program using the following data ; confidence interval 95% , power of test 80% , ratio of unexposed/exposed 1, percent of patients with successful management of acute perforated peptic ulcer by surgical intervention 90% and those with successful management by endoscopy 99% , odds ratio 99%, and risk ratio 2 , so the calculated sample size equal 100 patients divided into two equal groups. Group (1) included 50 patients managed by combined endoscopic & radiologic intervention , group (2) included 50 patients managed by surgery.

DETAILED DESCRIPTION:
The investigators included all patients who were developed acute perforated peptic ulcer manifestations and were admitted to our hospital between December 2019 to August 2021. The study was approved by the research and Ethics committee of our university and performed in accordance with the code of ethics of the world medical association (Declaration of Helsinki) for studies involving humans. A written informed consent was obtained from all participants. The sample size was calculated using open Epi program using the following data ; confidence interval 95% , power of test 80% , ratio of unexposed/exposed 1, percent of patients with successful management of acute perforated peptic ulcer by surgical intervention 90% and those with successful management by endoscopy 99% , odds ratio 99%, and risk ratio 2 , so the calculated sample size equal 100 patients divided into two equal groups. Group (1) included 50 patients managed by combined endoscopic & radiologic intervention , group (2) included 50 patients managed by surgery. Any patients with acute perforated peptic ulcer manifestations and age over 18 years were included. Patients presented with septic shock and age below 18 years were excluded.

Perioperative measures:

In this prospective randomized controlled trial , all patients were subjected to the followings: patients were selected by randomization method , Full history taking , Complete physical examination , laboratory investigations ( complete blood picture , liver and kidney functions , coagulation profile ) , radiological investigations ( chest x- ray erect , abdominal & pelvic u/s ).

Surgical techniques :

Traditional surgical exploration and Graham omental patch repair with abdominal lavage either open or laparoscopy was done for group (2). For group (1) endoscopic management using stent , clipping and sewing combined with radiologic interventional drainage was used. For duodenal ulcer only metallic stent was used due to narrow space while for gastric ulcer either stent , clipping and sewing were used due to capacious space.

Metallic stent:

Upper GI endoscopy ( Model GIF - 2TH180; Olympus , Tokyo, Japan) was done , allowing through it stent placement. The endoscopy was passed beyond the site of perforation , a guide wire was passed through the endoscopy into the proximal part of the jejunum and a partially covered duodenal stent ( Hanaro, MI-tech Korea) was advanced and released over the wire ( Jagwire ; Boston Scientific , Marlborough , M , USA) to cover the perforation site. Attention was taken to place the oral part of the stent above the pylorus and the covered part of the stent at site of perforation.

At same time of stent placement a radiologic interventional team worked and drainage was done & 2 intra-peritoneal tube drains were inserted one was placed sub-hepatic another was placed in the pelvis.

During postoperative day one a methylene blue test was done . and blue color was observed in the drain.

Stent was removed 3 weeks later and site of perforation was observed . if there was any sings of remaining perforation a new stent was placed for another 3 weeks.

Endoscopic clips:

Clips are used to approximate the tissue surrounding the defect to effect closure. Standard clips should be deployed perpendicular to the long axis of the defect. If needed, multiple clips can be placed sequentially, starting at either edge of a defect and meeting at the center. Currently available through-the-scope clips achieve superficial tissue apposition engaging the mucosa and submucosa (with 1.2-mm-wide and 6-mm-long arms capable of an approximately 12-mm grasp), and have been used in conjunction with thermal ablation or mechanical scraping of the tissue around the edges of the defect to achieve a more resilient seal. The Over-the-Scope Clip (Ovesco Endoscopic AG, Tubingen, Germany) is a nitinol clip placed on a cap at the endoscope tip . Unlike clips inserted through the endoscope, the OVESCO can perform full-thickness apposition.

At same time a radiologic interventional team worked and drainage was done & 2 intra-peritoneal tube drains were inserted one was placed sub-hepatic another was placed in the pelvis.

During postoperative day one a methylene blue test was done . and blue color was observed in the drain.

Sewing:

The Stomaphy X suturing system (Endo Gastric Solutions, Redmond, WA) and the Apollo Over Stitch (Apollo Endo surgery, Austin, TX), which creates full-thickness plications , has shown early success .

At same time a radiologic interventional team worked and drainage was done & 2 intra-peritoneal tube drains were inserted one was placed sub-hepatic another was placed in the pelvis.

During postoperative day one a methylene blue test was done . and blue color was observed in the drain.

Follow up after surgery and discharge from the hospital:

The investigators examined the patients clinically, made routine laboratory investigations , and for group (1) upper GI endoscopy at 2 weeks later.

Statistical analysis:

The collected data were analyzed by computer using Statistical Package of Social Services version 22 (SPSS), Data were represented in tables and graphs, Continuous Quantitative variables e.g. age were expressed as the mean ± SD & (range), and categorical qualitative variables were expressed as absolute frequencies (number) & relative frequencies (percentage).

Suitable statistical tests of significance were used after checked for normality. Categorical data were cross tabulated and analyzed by the Chi-square test or Fisher's Exact Test; Continuous data were evaluated by student t- test. The results were considered statistically significant when the significant probability was less than 0.05 (P < 0.05). P-value < 0.001 was considered highly statistically significant (HS), and P-value ≥ 0.05 was considered statistically insignificant (NS).

ELIGIBILITY:
Inclusion Criteria:

* Any patients with acute perforated peptic ulcer manifestations . _ age over 18 years.

Exclusion Criteria:

* Patients presented with septic shock . _ age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
incidence of complications after combined endoscopic & radiologic intervention | within one week after the endoscopy
  incidence of complications after combined endoscopic & radiologic intervention

SECONDARY OUTCOMES:
incidence of mortality after combined endoscopic & radiologic intervention | within one month after the endoscopy
  incidence of mortality after combined endoscopic & radiologic intervention

CONTACTS AND LOCATIONS:
Overall Officials: Said Mohamed Negm, MD, Principal Investigator — ZAGAZIG UNIVERSITY HOSPITALS
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqua, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Negm S, Mohamed H, Shafiq A, AbdelKader T, Ismail A, Yassin M, Mousa B, Abozaid M, Orban YA, Al Alawi M, Farag A. Combined endoscopic and radiologic intervention for management of acute perforated peptic ulcer: a randomized controlled trial. World J Emerg Surg. 2022 May 24;17(1):24. doi: 10.1186/s13017-022-00429-9. PMID 35610657